CLINICAL TRIAL: NCT04028713
Title: A Non-inferiority Study on Dose Reduction of Adalimumab in Psoriasis Patients
Brief Title: Dose Tapering Study of Adalimumab in Psoriasis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Too slow inclusion rate.
Sponsor: University Hospital, Ghent (Other)
Collaborators: KU Leuven (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC-03439
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis Vulgaris
Keywords: Therapeutic drug monitoring; Psoriasis; Adalimumab
MeSH Terms: conditions — Psoriasis | interventions — Dried Blood Spot Testing; Drug Tapering

STUDY DESIGN:
Intervention Model Description: A randomized non-inferiority study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dosing group (Active Comparator): Patients will continue to receive adalimumab according to the standard dosing schedule.
  Interventions: Procedure: Venapuncture; Procedure: Dried blood spot
- Dose tapering group (Experimental): Adalimumab dosing frequency will be lowered in patients who have supratherapeutic serum trough levels of adalimumab.
  Interventions: Procedure: Venapuncture; Procedure: Dried blood spot; Drug: Dose reduction

INTERVENTIONS:
Procedure: Venapuncture — Blood samples will be collected to determine the serum trough levels and anti-drug antibodies of adalimumab.
Procedure: Dried blood spot — A subset of patients will sample additionally by using the dried blood sampling technique.
Drug: Dose reduction — Adalimumab dosing frequency will be lowered in patients who have supratherapeutic serum trough levels of adalimumab.
  Arms: Dose tapering group

SUMMARY:
The optimal therapeutic serum trough level (Ctrough) of adalimumab was defined between 3,5 and 7,0 µg/ml in patients with plaque type psoriasis. An adalimumab Ctrough above this therapeutic range did not add clinical response. Based on this therapeutic window, the introduction of dose adjustments based on Ctroughs (therapeutic drug monitoring) will be further validated in a prospective randomized-controlled trial. Here, we aim to determine whether, in patients with a good clinical response and supratherapeutic adalimumab Ctroughs, dose reduction is able to maintain favorable clinical outcome.

DETAILED DESCRIPTION:
Patients will be included after signing informed consent and randomized in either a standard dose arm or a concentration based arm based on prior Ctrough measurements. In the concentration based arm, dosing frequency will be lowered to once every 3 weeks. If patients still have supratherapeutic Ctroughs of adalimumab, these patients will continue adalimumab self-administration every 4 weeks. In the standard based arm, patients will continue on standard dosing schedule. During each study visit blood will be taken in order to quantify Ctroughs. In addition, Psoriasis Area and Severity Index (PASI) and Investigator's Global Assessment (IGA) score will be evaluated by a physician. Patients complete the Dermatology Life Quality Index (DLQI) and European quality of life EQ-5D instrument at each visit. In addition, in a subset of patients in each treatment arm, additional sampling will be collected by dried blood spot sampling in order to build a PK(PD) model for adalimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a clinical or histological diagnosis of chronic plaque-type psoriasis for at least 6 months prior to inclusion
2. Participants must have a stable disease during maintenance on adalimumab (absolute PASI < 3)
3. Participants are not allowed to use topical steroids from 7 days before randomization until the end of the study (week 48).
4. Participants must sign an ICF indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

1. Participants who have currently a predominant nonplaque form of psoriasis
2. Participants who are pregnant, nursing or planning a pregnancy while enrolled in the study or within 12 weeks after receiving the last administration of study intervention
3. Participants who are unable or unwilling to undergo multiple venapunctures
4. Participants who are treated according to a different dosing schedule than standard dosing of adalimumab (regular dose regimen every 2 weeks; 40 mg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Clinical response | Week 0- Week 48
  The proportion of patients in each group in clinical remission (absolute PASI < 2) at year 1 after optimization

SECONDARY OUTCOMES:
The proportion of patients in each group with serum trough levels of adalimumab within the optimal interval. | Week 0- Week 48
The proportion of patients in each group with anti-drug antibodies (ADA) against adalimumab. | Week 0- Week 48
Relapse | Week 0- Week 48
  The proportion of patients in each group who relapses (defined as the need for dose escalation (not in the standard based dosing arm))

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof, dr, Principal Investigator — University Hospital, Ghent
Locations (7):
- Belgium (7):
  - AZ Maria Middelares, Ghent, East-Flanders
  - AZ Sint-Lucas, Ghent, East-Flanders
  - University Hospital Ghent, Ghent, East-Flanders
  - Private practice Dermatology, Maldegem, East-Flanders
  - University Hospital Leuven, Leuven, Vlaams-Brabant
  - AZ Delta Rembert, Torhout, West-Flanders
  - AZ Sint-Jan, Bruges, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soenen R, Stove C, Capobianco A, De Schutter H, Dobbelaere M, Mahjor T, Follens M, Lambert J, Grine L. Promising Tools to Facilitate the Implementation of TDM of Biologics in Clinical Practice. J Clin Med. 2022 May 26;11(11):3011. doi: 10.3390/jcm11113011. PMID 35683398
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35683398/